CLINICAL TRIAL: NCT02360488
Title: Telerehabilitation in the Home Versus Therapy In-Clinic for Patients With Stroke An Assessor-blind, Randomized, Non-inferiority Trial
Brief Title: Telerehabilitation in the Home Versus Therapy In-Clinic for Patients With Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Steven C. Cramer, MD, Professor of Neurology and Anatomy & Neurobiology; Vice Chair for Research in the Dept. Neurology, Clinical Director of the Stem Cell Research Center, Associate Director of the UC Irvine CTSA (Institute for Clinical & Translational Science), University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1U01NS091951-01A1 (NIH)
Record Dates: First submitted 2015-02-05; First posted 2015-02-10 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telerehabilitation Therapy (Experimental): The Telerehabilitation arm of this study will deliver rehabilitation treatment sessions via an in-home internet-connected computer. A major component of the system is the use of games to promote therapeutically relevant movements. The subject will perform daily assigned home-based telerehabilitation games and exercises and 5 minutes of stroke education, all guided by the telerehabilitation system.During half of the sessions, therapists will initiate a videoconference with the subject's telerehabilitation system to discuss progress, issues, and revise treatment plans as needed.
  Interventions: Device: Telerehabilitation Therapy
- In-Clinic Therapy (Active Comparator): The in-clinic arm of this study will deliver half of the rehabilitation treatment sessions at a study site providing traditional outpatient therapy, continuously supervised by a licensed therapist. The unsupervised therapy sessions will take place in the patient's home, and will be guided by an individualized booklet generated and printed by the Treatment Therapist and distributed to the subject during the first in-clinic therapy visit. The content of the unsupervised therapy sessions will be matched to the same exercise and training components provided during the subject's in-clinic supervised therapy sessions. In addition, at the start of each of the unsupervised sessions, all subjects will receive 5 minutes of stroke education.
  Interventions: Behavioral: In-Clinic Therapy

INTERVENTIONS:
Device: Telerehabilitation Therapy — 18 days of supervised sessions via videoconference and 18 days of unsupervised sessions.
  Arms: Telerehabilitation Therapy
Behavioral: In-Clinic Therapy — 18 days of therapist supervised sessions and 18 days of unsupervised in home sessions.
  Arms: In-Clinic Therapy

SUMMARY:
The current study will test the effectiveness of a novel home-based telehealth system designed to improve motor recovery and patient education after stroke. A total of 124 subjects (the number may be larger depending on the rate of subject dropout) with arm motor deficits 4-36 weeks after a stroke due to ischemia or to intracerebral hemorrhage will be randomized to receive 6 weeks of intensive arm motor therapy (a) in a traditional in-clinic setting or (b) via in-home telerehabilitation (rehabilitation services delivered to the subject's home via an internet-connected computer). The intensity, duration, and frequency of this therapy will be identical across the two groups, with subjects in both treatment arms receiving 36 sessions (18 supervised and 18 unsupervised), 80 minutes each (including a 10 minute break), over 6 weeks. The primary endpoint is within-subject change in the arm motor Fugl-Meyer (FM) score from the Baseline Visit to 30 Day Follow-Up Visit. Arm motor status is the focus here because it is commonly affected by stroke, is of central importance to many human functions, and is strongly linked to disability and well being after stroke.

DETAILED DESCRIPTION:
Substantial evidence indicates that occupational and physical therapy improves outcomes after stroke, and that larger doses are associated with superior outcomes. However, many patients receive suboptimal doses of therapy for reasons that include cost, access, and difficulty with travel. This problem is likely to increase with time given the aging of the population and the increased rate with which patients survive stroke. Telehealth, defined as the delivery of health-related services and information via telecommunication technologies, has enormous potential to address this unmet need.

The current study will test the effectiveness of a novel home-based telehealth system designed to improve motor recovery and patient education after stroke. A total of 124 subjects (the number may be larger depending on the rate of subject dropout) with arm motor deficits 4-36 weeks after a stroke due to ischemia or to intracerebral hemorrhage will be randomized to receive 6 weeks of intensive arm motor therapy (a) in a traditional in-clinic setting or (b) via in-home telerehabilitation (rehabilitation services delivered to the subject's home via an internet-connected computer). The intensity, duration, and frequency of this therapy will be identical across the two groups, with subjects in both treatment arms receiving 36 sessions (18 supervised and 18 unsupervised), 80 minutes each (including a 10 minute break), over 6 weeks. The primary endpoint is within-subject change in the arm motor Fugl-Meyer (FM) score from the Baseline Visit to 30 Day Follow-Up Visit. Arm motor status is the focus here because it is commonly affected by stroke, is of central importance to many human functions, and is strongly linked to disability and well being after stroke.

Telerehabilitation will be evaluated using an assessor-blind, randomized, non-inferiority study design. This study seeks to establish comparable efficacy between the two treatment arms based upon a non-inferiority margin of 2.05 points on the arm motor Fugl-Meyer scale. Key study features include enrollment of a diverse stroke population, standardized and blinded outcomes assessment, a standardized treatment protocol, covariate-adaptive randomization, and use of an active comparator that is matched for duration, frequency, and intensity of therapy. The FDA has determined that this investigation is a non-significant risk device study.

A minimum of 5 clinical sites will participate in this study. Each clinical site will conduct all testing and treatment at a single central site, although each clinical site is encouraged to recruit subjects from their referral hospitals. At the central study site, an Assessment Therapist will perform all study testing, blinded to treatment assignment (the subject by necessity is not blinded), while a Treatment Therapist will provide in-clinic therapy as well as direct home-based telerehabilitation. Potential enrollees may be identified through any of several routes, for example, during the acute stroke admission at the clinical site or a referral hospital, during inpatient rehabilitation at the clinical site or a referral hospital, or through other means of community-based recruitment. Study conduct will be highly standardized, including selecting therapy content, delivering therapy, and testing.

The current study aims to critically evaluate the utility of a telehealth approach to motor therapy and stroke education. Telehealth has enormous potential to address unmet needs in the growing population of stroke survivors.

ELIGIBILITY:
Inclusion criteria

1. Age ≥18 years at the time of randomization
2. Stroke that is radiologically verified, due to ischemia or to intracerebral hemorrhage, and with time of stroke onset 4-36 weeks prior to randomization
3. Arm motor FM score of 22-56 (out of 66) at both the Screening Visit and Baseline Visit
4. Box & Block Test score with affected arm is at least 3 blocks in 60 seconds at the Screening Visit
5. Informed consent signed by the subject
6. Behavioral contract signed by the subject

Exclusion criteria

1. A major, active, coexistent neurological or psychiatric disease, including alcoholism or dementia
2. A diagnosis (apart from the index stroke) that substantially affects paretic arm function
3. A major medical disorder that substantially reduces the likelihood that a subject will be able to comply with all study procedures
4. Severe depression, defined as GDS Score >10
5. Significant cognitive impairment, defined as Montreal Cognitive Assessment score < 22
6. Deficits in communication that interfere with reasonable study participation
7. A new symptomatic stroke has occurred since the index stroke that occurred 4-36 weeks prior to randomization
8. Lacking visual acuity, with or without corrective lens, of 20/40 or better in at least one eye
9. Life expectancy < 6 months
10. Pregnant
11. Receipt of Botox to arms, legs, or trunk in the preceding 6 months, or expectation that Botox will be administered to the arm, leg, or trunk prior to completion of the 30 Day Follow Up Visit
12. Unable to successfully perform all 3 of the rehabilitation exercise test examples
13. Unable or unwilling to perform study procedures/therapy, or expectation of non-compliance with study procedures/therapy
14. Concurrent enrollment in another investigational study
15. Non-English speaking, such that subject does not speak sufficient English to comply with study procedures
16. Expectation that subject cannot participate in study visits
17. Expectation that subject will not have a single domicile address during the 6 weeks of therapy, within 25 miles of the central study site and with Verizon wireless reception.**

    * A site may enroll a person who does not meet exclusion criterion # 17 if this is specifically approved by the site's study PI.
    * Because Montreal Cognitive Assessment scores may be difficult to interpret for patients with aphasia, at the discretion of the site's study PI, exclusion criterion #5 ("MoCA score cannot be <22") can be waived.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-09; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven C Cramer, MD, Principal Investigator — University of California, Irvine
Locations (12):
- United States (12):
  - University of California, Irvine, Irvine, California
  - UCSD Stroke Center, San Diego, California
  - Brooks Rehabilitation Clinical Research Center, Jacksonville, Florida
  - Emory Rehabilitation Hospital, Atlanta, Georgia
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Spaulding Rehabilitation Hospital, Charlestown, Massachusetts
  - Kessler Institute for Rehabilitation, Saddle Brook, New Jersey
  - Mount Sinai, New York, New York
  - Burke Rehabilitation Hospital, White Plains, New York
  - MetroHealth Rehabilitation Institute of Ohio, Cleveland, Ohio
  - MUSC Center for Rehabilitation Research in Neurological Conditions, Charleston, South Carolina
  - Harborview Medical Center, Seattle, Washington

REFERENCES:
- [Background] Cramer SC, Sur M, Dobkin BH, O'Brien C, Sanger TD, Trojanowski JQ, Rumsey JM, Hicks R, Cameron J, Chen D, Chen WG, Cohen LG, deCharms C, Duffy CJ, Eden GF, Fetz EE, Filart R, Freund M, Grant SJ, Haber S, Kalivas PW, Kolb B, Kramer AF, Lynch M, Mayberg HS, McQuillen PS, Nitkin R, Pascual-Leone A, Reuter-Lorenz P, Schiff N, Sharma A, Shekim L, Stryker M, Sullivan EV, Vinogradov S. Harnessing neuroplasticity for clinical applications. Brain. 2011 Jun;134(Pt 6):1591-609. doi: 10.1093/brain/awr039. Epub 2011 Apr 10. PMID 21482550
- [Background] Kleim JA, Jones TA. Principles of experience-dependent neural plasticity: implications for rehabilitation after brain damage. J Speech Lang Hear Res. 2008 Feb;51(1):S225-39. doi: 10.1044/1092-4388(2008/018). PMID 18230848
- [Background] Kwakkel G, Wagenaar RC, Twisk JW, Lankhorst GJ, Koetsier JC. Intensity of leg and arm training after primary middle-cerebral-artery stroke: a randomised trial. Lancet. 1999 Jul 17;354(9174):191-6. doi: 10.1016/S0140-6736(98)09477-X. PMID 10421300
- [Background] Langhorne P, Coupar F, Pollock A. Motor recovery after stroke: a systematic review. Lancet Neurol. 2009 Aug;8(8):741-54. doi: 10.1016/S1474-4422(09)70150-4. PMID 19608100
- [Background] Brennan DM, Tindall L, Theodoros D, Brown J, Campbell M, Christiana D, Smith D, Cason J, Lee A; American Telemedicine Association. A blueprint for telerehabilitation guidelines--October 2010. Telemed J E Health. 2011 Oct;17(8):662-5. doi: 10.1089/tmj.2011.0036. Epub 2011 Jul 26. No abstract available. PMID 21790271
- [Derived] Cramer SC, Le V, Saver JL, Dodakian L, See J, Augsburger R, McKenzie A, Zhou RJ, Chiu NL, Heckhausen J, Cassidy JM, Scacchi W, Smith MT, Barrett AM, Knutson J, Edwards D, Putrino D, Agrawal K, Ngo K, Roth EJ, Tirschwell DL, Woodbury ML, Zafonte R, Zhao W, Spilker J, Wolf SL, Broderick JP, Janis S. Intense Arm Rehabilitation Therapy Improves the Modified Rankin Scale Score: Association Between Gains in Impairment and Function. Neurology. 2021 Apr 6;96(14):e1812-e1822. doi: 10.1212/WNL.0000000000011667. Epub 2021 Feb 15. PMID 33589538
- [Derived] Cramer SC, Dodakian L, Le V, See J, Augsburger R, McKenzie A, Zhou RJ, Chiu NL, Heckhausen J, Cassidy JM, Scacchi W, Smith MT, Barrett AM, Knutson J, Edwards D, Putrino D, Agrawal K, Ngo K, Roth EJ, Tirschwell DL, Woodbury ML, Zafonte R, Zhao W, Spilker J, Wolf SL, Broderick JP, Janis S; National Institutes of Health StrokeNet Telerehab Investigators. Efficacy of Home-Based Telerehabilitation vs In-Clinic Therapy for Adults After Stroke: A Randomized Clinical Trial. JAMA Neurol. 2019 Sep 1;76(9):1079-1087. doi: 10.1001/jamaneurol.2019.1604. PMID 31233135

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telerehabilitation Therapy | In-Clinic Therapy
Started | 62 | 62
Completed | 59 | 55
Not Completed | 3 | 7

BASELINE CHARACTERISTICS:
Population: All subjects who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Telerehabilitation Therapy | In-Clinic Therapy | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (14) | 60 (13) | 61 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 20 | 34
  Male | 48 | 42 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 59 | 62 | 121
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 18 | 33
  White | 41 | 39 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 62 | 62 | 124
Arm motor Fugl-Meyer score [Mean (Standard Deviation); unit: units on a scale] — The full name of this scale is the arm motor Fugl-Meyer scale. it measures arm motor impairment, which is in the body structure/function domain. It consists of 33 individual assessments that are summed to generate a total arm motor Fugl-Meyer score. Scores range from 0-66, which higher values being better (and so 66 being normal). There are no subscores evaluated.
  units on a scale | 42.8 (7.8) | 42.7 (8.7) | 42.8 (8.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Arm Motor Fugl-Meyer Score From Baseline to 30 Days Post-therapy
Description: The full name of this scale is the arm motor Fugl-Meyer scale. it measures arm motor impairment, which is in the body structure/function domain. It consists of 33 individual assessments that are summed to generate a total arm motor Fugl-Meyer score. Scores range from 0-66, which higher values being better (and so 66 being normal). There are no subscores evaluated.
Time Frame: from the Baseline Visit to the 30 Day Follow Up Visit
Population: Intention-to-Treat with multiple imputation of missing outcomes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telerehabilitation Therapy | In-Clinic Therapy
Number analyzed (Participants) | 62 | 62
units on a scale | 7.86 (6.68) | 8.36 (7.04)
Statistical Analysis 1: Comparison: Telerehabilitation Therapy vs In-Clinic Therapy; Test type: Non-Inferiority — The trial aimed to establish comparable efficacy based upon a non-inferiority margin of 30% of the change in Fugl-Meyer score in the In-Clinic group. Under these assumptions at alpha=0.05 and assuming SD=3.8 points, 124 subjects would need to be enrolled to provide 85% power; this sample was pursued independent of subject dropouts; p = .96, Regression, Linear; The model was adjusted for study site, age, time post-stroke, stroke subtype, and baseline Fugl-Meyer score; Mean Difference (Net) = 0.06, 95% CI 2-sided [-2.14 to 2.26]

ADVERSE EVENTS:
Time Frame: Baseline to 30 days post-therapy
Description: Adverse events were collected, and those possibly or probably reasonably/definitely related to study procedures are reported.
Arm/Group | Telerehabilitation Therapy | In-Clinic Therapy
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62
Serious Adverse Events (participants affected / at risk) | 1/62 | 6/62
Other Adverse Events (participants affected / at risk) | 10/62 | 7/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telerehabilitation Therapy (N=62) | In-Clinic Therapy (N=62)
Dizziness (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Fall (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Limb fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Subdural hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telerehabilitation Therapy (N=62) | In-Clinic Therapy (N=62)
Arm/shoulder pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 4 (4)
Fatigue (Nervous system disorders) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-04-21): https://cdn.clinicaltrials.gov/large-docs/88/NCT02360488/Prot_SAP_ICF_000.pdf